CLINICAL TRIAL: NCT04663477
Title: Patient-Completed Caprini Risk Score for Venous Thromboembolism Risk Assessment Developed and Validated From 1017 Medical and Surgical Patients: a Diagnostic Study
Brief Title: Development and Validation of the Patient-completed Caprini Risk Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Deputy Director of the Second Department of Respiratory and Critical Care Medicine in China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: VTE-CRS-study
Record Dates: First submitted 2020-11-28; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Venous Thromboembolism
Keywords: VTE risk; Caprini; Patient-complete; Validation
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trained nurse-completed CRS
  Interventions: Diagnostic Test: patient-completed Caprini Risk Score
- Patient-completed CRS
  Interventions: Diagnostic Test: patient-completed Caprini Risk Score

INTERVENTIONS:
Diagnostic Test: patient-completed Caprini Risk Score — The participants will be asked to complete patient-completed Caprini Risk Score

SUMMARY:
The investigators aimed to test the reliability and validity of the Chinese version of patient-completed CRS in hospitalized patients and to evaluate whether this form can be widely used in clinical practice instead of only health care workers' evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* patients with first admission to the medical and surgical units within 24 hours
* willingness to participate in the study

Exclusion Criteria:

* patients with a diagnosis of PTE or DVT on admission
* patients with cognitive impairment
* inability to read or write
* patients with mental diseases
* patients with visual impairment
* refusal to cooperate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will recruite nearly 500 inpatients from the surgical unit and nearly 500 inpatients from the medical unit between January 1 and December 31, 2019
Sampling Method: Probability Sample
Enrollment: 1017 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Question-to-question agreement between patient-completed and nurse-completed CRS | one year
  The investigators will use kappa value to compare the question-to-question agreement level between nurse and patient-completed Caprini Risk Score

SECONDARY OUTCOMES:
Correlation and difference between the scores calculated by patient-completed and nurse-completed CRS | one year
  The Spearman correlation coefficient was used to measure the correlation and difference between patient-completed and nurse-completed CRS.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Frendship hospital, Beijing, China